CLINICAL TRIAL: NCT05970159
Title: The Impacts of preopeRative sErum Albumin Levels on Postoperative Outcomes in Chinese HCC Patients Treated With Surgical Operation: REAL Study
Brief Title: Impact of Preoperative Serum Albumin Level on Postoperative Outcomes in Chinese HCC Patients Treated With Surgery
Acronym: REAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: B2023-216
Record Dates: First submitted 2023-07-18; First posted 2023-08-01 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Albumin; Hepatectomy; Liver transplantation; Postoperative outcomes
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypoalbuminemia group: Patients with hepatocellular carcinoma whose preoperative serum albumin concentration are < 36g/L.
- Normal group: Patients with hepatocellular carcinoma whose preoperative serum albumin concentration are ≥ 36g/L.

SUMMARY:
This is an observational and retrospective cohort study to evaluate the impact of the preoperative serum albumin concentration on postoperative outcomes among hepatocellular carcinoma (HCC) patients who received hepatectomy or liver transplantation.

DETAILED DESCRIPTION:
The impact of hypoalbuminemia on postoperative outcomes has been the subject of several investigations which agreed that hypoalbuminemia is an important risk factor for mortality and morbidity after various types of surgical operations. Unfortunately, there are limited real-world data to establish the correlation between hypoalbuminemia and hepatectomy or liver transplantation postoperative complications in China. This study will evaluate the impact of the preoperative serum albumin concentration on postoperative outcomes among hepatocellular carcinoma (HCC) patients who received hepatectomy or liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed with HCC confirmed by histology/cytology or clinically criteria regardless of gender.
* HCC Patients who had received the first hepatectomy or liver transplantation (LT).
* Age ≥18 years at the start date of the hepatectomy or LT.
* HCC patients who had the value of serum albumin within 7 days prior to the surgery.
* HCC patients who had exemption of informed consent.

Exclusion Criteria:

* HCC Patients with extrahepatic metastasis or other malignant tumours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who met the criteria for inclusion in this real-world study from Zhongshan Hospital, Fudan University will be included. According to a preliminary feasibility department investigation, a sample size of approximately 480 subjects will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | up to 2 weeks
  Complications following surgery that occurred during hospitalization. For the hepatectomy cohort of patients, postoperative complications included incision, urinary tract and abdominal infections, pleural fluid, ascites, post-hepatectomy hemorrhage bile leakage, post hepatectomy liver failure, renal insufficiency, multiple organ dysfunction syndrome, pneumonia and pulmonary embolism, etc. For the LT cohort of patients, postoperative complications included primary nonfunction, hemorrhage, hepatic artery thrombosis, hepatic vein thrombosis, bile leakage, acute kidney injury, deep wound infections and catheter-related infections.

SECONDARY OUTCOMES:
Mortality | up to 2 weeks
  Death occurring during the postoperative hospital stay.

OTHER OUTCOMES:
Days of hospital stay | up to 2 weeks
  The length of stay in hospital after surgery.
Days of ICU stay | up to 4 weeks
  The length of stay in ICU after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Huichuan Sun, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ma KW, Cheung TT, She WH, Chok KSH, Chan ACY, Dai WC, Lo CM. Risk prediction model for major complication after hepatectomy for malignant tumour - A validated scoring system from a university center. Surg Oncol. 2017 Dec;26(4):446-452. doi: 10.1016/j.suronc.2017.08.007. Epub 2017 Sep 9. PMID 29113664
- [Result] Poon RT, Fan ST, Lo CM, Liu CL, Lam CM, Yuen WK, Yeung C, Wong J. Improving perioperative outcome expands the role of hepatectomy in management of benign and malignant hepatobiliary diseases: analysis of 1222 consecutive patients from a prospective database. Ann Surg. 2004 Oct;240(4):698-708; discussion 708-10. doi: 10.1097/01.sla.0000141195.66155.0c. PMID 15383797